CLINICAL TRIAL: NCT03636516
Title: Effect of Double J Stent on Outcomes of Extracorporeal Shock Wave Lithotripsy Treatment of Moderate Sized Renal Pelvic Stones: A Randomized Prospective Study
Brief Title: Effect of Double J Stent on Outcomes of Extracorporeal Shock Wave Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Akif Erbin, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456789
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- jj stent yes (Active Comparator)
  Interventions: Device: SWL
- jj stent no (Active Comparator)
  Interventions: Device: SWL

INTERVENTIONS:
Device: SWL — extracorporeal shockwave lithotripsy apply

SUMMARY:
Background: Many studies showed that stone-free rates (SFRs) after extracorporeal shock wave lithotripsy (SWL) might be related to both the patient (body mass index; BMI, skin-to-stone distance; SSD), and stone related factors (location, stone size, and stone density). However, the possible effect of pre-stenting on success as well as complication rates after SWL has not been evaluated in detail to date. Taking this fact into account, the effect of pre-stenting on the outcomes of SWL treatment in renal stones must be evaluated in the absence of possible effects induced by the patient and stone-related factors. Aim: To evaluate the effect of double J (JJ) stents on SWL treatment of moderate sized (15-25-mm) renal pelvic stones. Study design: Randomized prospective study Methods: Between January 2016 and December 2017, a total of 152 adult patients who were planned to undergo SWL for a single radiopaque renal pelvic stone were included in the study. Patients with solitary kidney, congenital abnormality, skeletal tract abnormalities, previous urinary system surgery, hydronephrosis (grade 2 or more), untreated urinary tract infection, bleeding disorder, and suspected pregnancy were excluded. The remaining 114 patients were randomly divided into two groups; nonstented and stented. Twenty-two patients whose stone could not be fragmented despite 3 consecutive sessions were also excluded from the study. A total of 92 patients (54 non-stented and 38 stented) were included in the final analysis.

DETAILED DESCRIPTION:
Study design Between January 2016 and December 2017, a total of 152 adult (age > 18 years) patients who were planned to undergo extracorporeal shock wave lithotripsy (SWL) for a single radiopaque renal pelvic stone with a largest diameter of 15 to 25 mm were included in the study. Patients with solitary kidneys, congenital abnormalities, skeletal system abnormalities, previous urinary system surgery, hydronephrosis (grade 2 or more), untreated urinary tract infection, bleeding disorder, and suspected pregnancy were excluded from the study. The remaining 114 patients were randomly divided into two groups as non-stented (n=67) and stented (n=47). Randomization was performed by flipping a coin. During SWL procedures, 22 patients whose stone could not be fragmented despite 3 consecutive sessions were also excluded from the study. A total of 92 patients (54 non-stented and 38 stented) were included in the final analysis.

Preprocedural evaluation All patients were evaluated preoperatively using non-contrast computed tomography (CT). Prior to treatment, a complete urine test, if needed urine culture and antibiogram test, simple serum biochemistry and coagulation tests were performed in all patients. The impact of patient-related factors (age, sex, body mass index;BMI), stone-related factors (laterality, stone size and Hounsfield units; HU), renal parenchymal thickness (RPT), and skin-to-stone distance (SSD) on fragmentation were analyzed. Body mass index (BMI) was calculated by dividing the weight (kg) by the square of the height (m2). CT with 5-mm contiguous sections at 120 kw and 90 milliampere (mA) was performed in all patients using a multidetector row helical CT scanner (Somatom Plus; Siemens, Germany). The longitudinal stone dimension was calculated by multiplying collimation thickness and the number of images in which the stone seen. The transverse dimension was chosen as the diameter of stone from the image showing its largest width. The maximum dimension of the stone was accepted as the highest value measured, either the longitudinal or transverse diameter. The average CT attenuation value as the representative HU was measured by drawing a region of interest smaller than the stone in the image showing the stone in the largest dimension. The SSD was calculated by measuring the distance from the skin to the stone at posterolateral 45°. All patients signed an informed consent form for SWL and pre-stenting. Stent size was 4.8 French and 26 cm.

SWL technique SWL was performed with an electromagnetic lithotripter Compact Sigma (Dornier Med Tech System Gesellschaft mit beschränkter Haftung; GmbH, Weßling, Germany) by the same operator, with the patient in the supine position, and with a standardized treatment angle under both fluoroscopic and ultrasonic guidance. SWL procedures were performed with analgesic application (75 mg diclofenac sodium). If needed, a compression bag was used to decrease stone movement caused by respiration. Each session was completed either after application of a total of 3000 shock waves or when the stone was completely disintegrated. The degree of shock wave power delivered during SWL was recorded as 1 to 6 and the shock wave frequency was 90/minute. Individual power settings were adjusted according to the patient's tolerance. Patients were evaluated 1 week after each session through abdominal kidneys, ureters, and urinary bladder (KUB) X-ray and repeat treatment was performed in cases of inadequate disintegration. Management was stopped when there was no disintegration despite 3 SWL sessions. No patients received medical expulsive treatment (MET) before or after SWL sessions. JJ stents were removed after 4 weeks. In view of the radiographic assessment with CT performed 4 months following the last SWL session, treatment results were categorized as either successful or unsuccessful according to whether there were any residual stone fragments. During SWL sessions and after treatment, the number of emergency department visits and analgesic consumption were recorded.

Statistical analysis Data were analyzed using the Statistical Package for the Social Sciences software version 19 (SPSS Inc., Chicago, Illinois, USA). Descriptive statistics were determined for the mean, standard deviation, lowest and highest, and ratio values. The distribution of the variables was measured using the Kolmogorov-Smirnov test. Univariate (Chi-square or t-test) tests were performed to determine whether there was a statistically significant difference for characteristics between the stented and non-stented groups. If parameters did not show normal dispersion, the Mann-Whitney U test, which is the nonparametric equivalent of the t-test, was performed. The threshold for statistical significance was accepted as p < 0.05 for all analyses.

ELIGIBILITY:
Inclusion Criteria:Between January 2016 and December 2017, a total of 152 adult (age > 18 years) patients who were planned to undergo ESWL for a single radiopaque renal pelvic stone with a largest diameter of 15 to 25 mm were included in the study.

-

Exclusion Criteria:

* Patients with solitary kidneys, congenital abnormalities, skeletal system abnormalities, previous urinary system surgery, HN (grade 2 or more), untreated urinary tract infection, bleeding disorder, and suspected pregnancy were excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients, who have JJ stent or not, with successful SWL treatment. | 15 weeks
  Number of patients, who have JJ stent or not, with successful SWL treatment which assessed after 3 months following the last SWL session.

IPD SHARING:
Plan to Share IPD: No